CLINICAL TRIAL: NCT00097812
Title: A Study to Assess the Safety, Tolerability, and Efficacy of Switching Patients Currently on Oral Bisphosphonate to Zoledronic Acid
Brief Title: Switching Osteoporosis Patients Currently on Oral Bisphosphonate to Zoledronic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446H2313
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Osteoporosis
Keywords: osteoporosis, osteopenia, post-menopausal, zoledronic acid
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: zoledronic acid

SUMMARY:
The purpose of this study is to assess bone mineral density in patients switching from an oral bisphosphonate to zoledronic acid, compared to those staying on the oral bisphosphonate.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women between 45 and 79 years of age
* Must be osteopenic/osteoporotic
* Treatment with oral bisphosphonate for at least 1 year

Exclusion Criteria:

* Any woman of child bearing potential
* Treatment with other bone active agents

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 45 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To compare % change in Lumbar Spine BMD from Baseline to Month 12 in ZOL (annual i.v. infusion) vs Alendronate (weekly oral) osteoporotic post-menopausal women populations

SECONDARY OUTCOMES:
To compare Biomarkers of bone turnover in the annual Zol i.v. and weekly alendronate populations
To demonstrate continued bone remodeling by evaluation of bone biopsies in a subset of patients
To assess patient preferences for annual i.v. therapy compared to weekly oral therapy through a patient questionnaire

CONTACTS AND LOCATIONS:
Locations (13):
- United States (12):
  - The Permanente Medical Group, Santa Rosa, California
  - Colorado Center for Bone Research, Lakewood, Colorado
  - Florida Medical Research Institute, Gainsville, Florida
  - Radiant Research, Stuart, Florida
  - University of Kansas School of Medicine/ Division of Endocrinology, Kansas City, Kansas
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Creighton University Osteoporosis Research Center, Omaha, Nebraska
  - Oregon Osteoporosis Center, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Radiant Research, Wyomissing, Pennsylvania
  - Puget Sound Osteoporosis Center, Seattle, Washington
- Novartis, Nuremberg, Germany